CLINICAL TRIAL: NCT00035594
Title: A Double-Blind, Placebo-Controlled, Multicenter, Randomized Study Evaluating the Prophylactic Use of Pegfilgrastim on the Incidence of Febrile Neutropenia in Subjects With Advanced Breast Cancer Treated With Single Agent Docetaxel
Brief Title: Pegfilgrastim as Support to Advanced Breast Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20010144
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Neutropenia
Keywords: Breast cancer; Neutropenia; Chemotherapy
MeSH Terms: conditions — Neutropenia; Breast Neoplasms | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Breast cancer patients receiving docetaxel chemotherapy and placebo.
  Interventions: Drug: pegfilgrastim
- Pegfilgrastim (Experimental): Breast cancer patients receiving docetaxel chemotherapy and pegfilgrastim.
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim — Growth factor (GCSF) administered to promote neutrophil development post-chemotherapy.

SUMMARY:
Physicians are conducting a clinical trial for patients with advanced breast cancer. Breast cancer can be treated with chemotherapy which can affect the bone marrow, where blood cells are produced. Neutrophils are a type of white blood cells that fight infection and are produced in the bone marrow. If the neutrophil count becomes low due to chemotherapy, a potentially serious condition called neutropenia occurs. Neutropenia is serious because it can affect the body's ability to protect against many types of infections. Pegfilgrastim is an investigational drug being evaluated for its potential ability to increase the number of neutrophils. The purpose of this study is to determine the safety and effectiveness of pegfilgrastim in preventing neutropenia following chemotherapy in patients with advanced breast cancer.

ELIGIBILITY:
* Advanced breast cancer
* 18 years of age or older
* Patients who will be receiving Taxotere (docetaxel) chemotherapy

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 928
Dates: Start 2002-02; Primary Completion 2004-02 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects developing febrile neutropenia | Through 4 cycles

SECONDARY OUTCOMES:
Incidence of hospitalization and IV antiinfective use associated with FN; also chemotherapy planned dose on time | Through 4 cycles

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Vogel CL, Wojtukiewicz MZ, Carroll RR, Tjulandin SA, Barajas-Figueroa LJ, Wiens BL, Neumann TA, Schwartzberg LS. First and subsequent cycle use of pegfilgrastim prevents febrile neutropenia in patients with breast cancer: a multicenter, double-blind, placebo-controlled phase III study. J Clin Oncol. 2005 Feb 20;23(6):1178-84. doi: 10.1200/JCO.2005.09.102. PMID 15718314
- [Derived] Lyman GH, Reiner M, Morrow PK, Crawford J. The effect of filgrastim or pegfilgrastim on survival outcomes of patients with cancer receiving myelosuppressive chemotherapy. Ann Oncol. 2015 Jul;26(7):1452-8. doi: 10.1093/annonc/mdv174. Epub 2015 Apr 7. PMID 25851633
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20010144.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/